CLINICAL TRIAL: NCT04114006
Title: Initial Analysis of Wide-area Transepithelial Sampling for the Detection of Gastric Neoplasia
Brief Title: Novel Screening Modality for Early Gastric Cancer
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Douglas Morgan MD, Professor of Medicine, Director, Division of Gastroenterology/ Hepatology, University of Alabama at Birmingham
Other Study IDs: IRB00001470; NCT05028296 (obsolete NCT alias)
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer
Keywords: gastric intestinal metaplasia; gastric neoplasia
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Potential patients will be recruited at participating sites based on routine care with clinical indications for upper endoscopy. Following informed consent, patients will undergo their scheduled endoscopy with standard forceps biopsies along with the transepithelial brush samples. All samples, biopsy and brush samples, will be sent for pathology analysis, per standard clinical practice.

DETAILED DESCRIPTION:
Potential patients will be recruited at participating sites based on routine care with clinical indications for upper endoscopy. Following informed consent, patients will undergo their scheduled endoscopy with standard forceps biopsies along with the transepithelial brush samples. All samples, biopsy and brush samples, will be sent for histologic analysis, with planned study of the diagnostic yields of each method.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed of the investigational nature of this study and given verbal and written informed consent in accordance with local, U.S., and international guidelines.
* Both males and females at least 18 years.
* Patients with clinical indications for upper endoscopy

Exclusion Criteria:

* Patients should not have an advanced medical or psychiatric conditions which that may limit their ability to participate in the study, as judged by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for upper endoscopy (e.g. dyspepsia)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of the WATS approach versus standard gastric biopsy mapping | 1-3 Years
  To compare the diagnostic yield of the WATS approach versus standard gastric biopsy mapping (per the updated Sydney system).

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Morgan, MD, MPH, Principal Investigator — University of Alabama at Birmingham; Ricardo Dominguez, MD, Principal Investigator — Hospital de Occidente Honduras
Locations (1):
- Hospital de Occidente, Santa Rosa de Copán, Copán Department, Honduras

REFERENCES:
- [Background] Vennalaganti PR, Kaul V, Wang KK, Falk GW, Shaheen NJ, Infantolino A, Johnson DA, Eisen G, Gerson LB, Smith MS, Iyer PG, Lightdale CJ, Schnoll-Sussman F, Gupta N, Gross SA, Abrams J, Haber GB, Chuttani R, Pleskow DK, Kothari S, Goldblum JR, Zhang Y, Sharma P. Increased detection of Barrett's esophagus-associated neoplasia using wide-area trans-epithelial sampling: a multicenter, prospective, randomized trial. Gastrointest Endosc. 2018 Feb;87(2):348-355. doi: 10.1016/j.gie.2017.07.039. Epub 2017 Jul 27. PMID 28757316
- [Background] ASGE STANDARDS OF PRACTICE COMMITTEE; Qumseya B, Sultan S, Bain P, Jamil L, Jacobson B, Anandasabapathy S, Agrawal D, Buxbaum JL, Fishman DS, Gurudu SR, Jue TL, Kripalani S, Lee JK, Khashab MA, Naveed M, Thosani NC, Yang J, DeWitt J, Wani S; ASGE Standards of Practice Committee Chair. ASGE guideline on screening and surveillance of Barrett's esophagus. Gastrointest Endosc. 2019 Sep;90(3):335-359.e2. doi: 10.1016/j.gie.2019.05.012. No abstract available. PMID 31439127
- [Background] Banks M, Graham D, Jansen M, Gotoda T, Coda S, di Pietro M, Uedo N, Bhandari P, Pritchard DM, Kuipers EJ, Rodriguez-Justo M, Novelli MR, Ragunath K, Shepherd N, Dinis-Ribeiro M. British Society of Gastroenterology guidelines on the diagnosis and management of patients at risk of gastric adenocarcinoma. Gut. 2019 Sep;68(9):1545-1575. doi: 10.1136/gutjnl-2018-318126. Epub 2019 Jul 5. PMID 31278206